CLINICAL TRIAL: NCT01491945
Title: Prospective, Multicenter, Single Arm Safety and Effectiveness Trial of the Endologix Fenestrated Stent Graft System for the Endovascular Repair of Juxtarenal/Pararenal (JAA/PAA) Aneurysms
Brief Title: Safety and Effectiveness Trial of the Ventana Fenestrated Stent Graft System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endologix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-0004
Record Dates: First submitted 2011-10-20; First posted 2011-12-14 (Estimated); Results first posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-09

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: Abdominal aortic aneurysm; Renal stent; Juxtarenal; Pararenal; Endovascular
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Ventana Fenestrated Stent Graft System (Experimental): Ventana Fenestrated Stent Graft System
  Interventions: Device: Ventana Fenestrated Stent Graft System

INTERVENTIONS:
Device: Ventana Fenestrated Stent Graft System — The Ventana Fenestrated Stent Graft System consists of the following:
  bifurcated stent graft, Ventana fenestrated proximal extension stent graft, and Xpand renal stent grafts

SUMMARY:
The purpose of this trial is to determine if the Ventana Fenestrated Stent Graft System is safe and effective for the endovascular repair of juxtarenal or pararenal aortic aneurysms.

DETAILED DESCRIPTION:
Study Objectives The objective of protocol CP-0004 is to study the safety and effectiveness of the Endologix Fenestrated System in the endovascular treatment of patients with juxtarenal and/or pararenal aortic aneurysms.

Study Design This clinical study is a prospective, non-randomized, multicenter study. The first patient enrolled at each site is designated as a 'Roll-In' group patient. Subsequently, enrolled patients are designated as 'Trial' group patients for primary endpoint analysis.

Primary Endpoint The primary safety endpoint is defined as the incidence of Major Adverse Events‡ (MAEs) within 30 days. The primary study effectiveness endpoint is Treatment Success at 1-year. This is defined as procedural technical success and the absence of aneurysm rupture; conversion to open surgical repair; Type I endoleak after 30 days; Type III endoleak; clinically significant migration; aneurysm enlargement; or secondary intervention for resolution of endoleak, limb occlusion, migration, aneurysm sac expansion and/or a device defect.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years old;
* Informed consent understood and signed and patient agrees to all follow-up visits;
* Have aortic aneurysm with maximum diameter ≥5.5cm, or between 4.5 and 5.5cm and rapidly expanding (>0.5cm in six months), or >50% larger than the normal aortic diameter
* Anatomically eligible for the Bifurcated System per the FDA-approved indications for use (IFU) and for the Fenestrated Stent Graft System:

  * Adequate iliac/femoral access compatible with the required delivery systems
  * Non-aneurysmal infrarenal aortic neck <15mm in length;
  * Most caudal renal artery to aortoiliac bifurcation length ≥70mm
  * SMA to aortoiliac bifurcation length ≥90mm;
  * Proximal non-aneurysmal aortic neck below the SMA with: diameter 18 to 34 mm; length ≥15 mm; angle ≤60° to the aneurysm sac;
  * Angle ≤60° (clock face) between the SMA and CA
  * Renal arteries both distal to the SMA by ≤35mm, within 30mm of each other axially, with 4 to 8mm lumen diameter, and with clock face angle of 90° to 210° to each other .Common iliac artery distal fixation site with: distal fixation length ≥15 mm; ability to preserve at least one hypogastric artery; diameter ≥10 mm and ≤23 mm; angle ≤90° to the aortic bifurcation.
* The Endologix Fenestrated Proximal Extension Stent must have the ability to overlap the bifurcated stent graft by at least 3cm.
* Aortic diameter at the most caudal renal artery of 18 to 36mm

Exclusion Criteria:

* Life expectancy <2 years as judged by the investigator;
* Psychiatric or other condition that may interfere with the study;
* Participating in the enrollment or 30-day follow-up phase of another clinical study;
* Known allergy to any device component;
* Coagulopathy or uncontrolled bleeding disorder;
* Contraindication to contrast media or anticoagulants;
* Ruptured, leaking, or mycotic aneurysm;
* Aortic dissection
* Serum creatinine (S-Cr) level >2.0 mg/dL;
* Traumatic vascular injury;
* Active systemic or localized groin infection;
* Connective tissue disease (e.g., Marfan's Syndrome);
* Recent (within prior three months) cerebrovascular accident or myocardial infarction;
* Prior renal transplant;
* Length of either renal artery to be stented <13mm;
* Significant occlusive disease of either renal artery (>70% stenosis);
* An essential accessory renal artery;
* Indispensable inferior mesenteric artery;
* Aneurysmal disease of the descending thoracic aorta;
* Clinically significant mural thrombus circumferentially in the suprarenal segment;
* Prior iliac artery stent implanted that may interfere with delivery system introduction;
* Unsuitable vascular anatomy;
* Pregnancy (female patient of childbearing potential only)
* Existing renal stent;
* Pre-planned need for concomitant procedure (e.g. surgical conduit for vascular access, hypogastric artery embolization/coil, renal artery angioplasty)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2013-03-03 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2018-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel G Clair, MD, Principal Investigator — The Cleveland Clinic
Locations (22):
- United States (22):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Heart Institute, Phoenix, Arizona
  - John Muir Medical Center Concord, CA, Concord, California
  - UCLA Medical Center, Los Angeles, California
  - VA Gainesville, Gainesville, Florida
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - Baptist East Hospital, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - William Beaumont Hospital, Royal Oak, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - University of North Carolina, Chapel Hill, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania
  - Methodist Hospital, Houston, Texas
  - Harborview Medical Center, Seattle, Washington
  - Charleston Area Medical Center, Charleston, West Virginia
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Ventana Fenestrated Stent Graft System: Objective is to study the safety and effectiveness of the Endologix Fenestrated Stent Graft System in the endovascular treatment of patients with juxtarenal and/or pararenal aortic aneurysms. Subjects were treated with the Ventana Fenestrated system in this arm and The Ventana Fenestrated Stent Graft System consisted of the following:
  bifurcated stent graft, Ventana fenestrated proximal extension stent graft, and Xpand renal stent grafts.
Period: Overall Study
Arm/Group | Ventana Fenestrated Stent Graft System
Started | 76
Completed | 25
Not Completed | 51
Not completed — Death | 30
Not completed — Withdrwan/LTF | 16
Not completed — Conversion | 4
Not completed — Missed Visit | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ventana Fenestrated Stent Graft System
Number analyzed (Participants) | 76
Age, Continuous [Mean (Standard Deviation); unit: Years] | 74.6 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 59
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 76
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 76
Serum Creatinine [Mean (Standard Deviation); unit: mg/dL] | 1.1 (0.3)
ASA Class [Count of Participants; unit: Participants] — Measure Description: ASA (American society of anesthesiologists) classifications explained below:
  ASA I A normal healthy patient ASA II A patient with mild systemic disease ASA III A patient with severe systemic disease ASA IV A patient with severe systemic disease that is a constant threat to life ASA V A moribund patient who is not expected to survive without the operation ASA VI A declared brain-dead patient whose organs are being removed for donor purposes
  Participants
    ASA Class 1 | 1
    ASA Class 2 | 27
    ASA Class 3 | 38
    ASA Class 4 | 10
estimated Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73m^2] | 77.9 (30.1)
Ankle Brachial Index [Mean (Standard Deviation); unit: Ratio (percentage)] — The Ankle Brachial Index (ABI) is the systolic pressure at the ankle, divided by the systolic pressure at the arm
  Greater than 1.4 Calcification/Vessel Hardening 1.0-1.4 Normal 0.9-1.0 Acceptable 0.8-0.9 Some Arterial Disease 0.5-0.8 Moderate Arterial Disease Less than 0.5 Severe Arterial Disease
  Ratio (percentage)
    ABI Left | 1.0 (0.2)
    ABI RIght | 1.0 (0.2)
Aneurysm Shape [Count of Participants; unit: Participants]
  Fusiform | 69
  Saccular | 7
Aneurysm Sac Diameter [Mean (Standard Deviation); unit: centimeter] | 5.8 (0.8)
Aneurysm Diameter (mm) [Count of Participants; unit: Participants]
  <45 mm | 1
  >=45-54 mm | 28
  >=55-64 mm | 33
  >=65-74 mm | 12
  >=75-84 mm | 1
  >=85 mm | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety- Number of Major Adverse Events at 30 Days
Description: Major Adverse Events = all cause death; bowel ischemia; myocardial infarction; paraplegia; renal failure; respiratory complications of stroke; blood loss >1000cc
Time Frame: 30 Days
Measure: Number; unit: Events
Arm/Group | Ventana Fenestrated Stent Graft System
Number analyzed (Participants) | 76
Events
  All Cause Death | 2
  Bowel Ischemia | 3
  Myocardial Infarction | 2
  Paraplegia | 1
  Procedural Blood Loss | 5
  Renal Failure 1 - Temporary/Permanent Hemodialysis | 4
  Renal Failure 2 - Serum Creatine >0.5mg/dL | 3
  Respiratory Failure 1 - Pneumonia | 1
  Respiratory Failure 2 - Ventilator >24hr | 2
  Stroke | 0

2. Primary Outcome: Effectiveness
Description: 1. Treatment Success is defined as Procedural technical success and absence of aneurysm rupture, conversion to open repair, Type I endoleak after 30 days, Type III endoleak, clinically significant migration; aneurysm enlargement; or secondary intervention for resolution of endoleak, limb occlusion, migration, aneurysm sac expansion and/or a device defect.
  2. Procedural Technical Success is defined as a subject with successful implant.
  3. Clinically Significant Device Migration: Core Lab reported aortic stent graft movement >10mm
  4. Type I/III/IV Endoleak: Core Lab reported endoleak: between the endograft and the vessel either at the proximal attachment point (Type IA), or at the distal attachment point (Type IB), or between endograft components (Type III) or transgraft (Type IV).
  5. Type II Endoleak: Core Lab reported endoleak emanating from a patent collateral vessel (e.g., inferior mesenteric artery, lumbar artery).
Time Frame: 1 Year
Measure: Count of Participants; unit: Participants
Arm/Group | Ventana Fenestrated Stent Graft System
Number analyzed (Participants) | 76
Participants
  Aneurysm Rupture | 0
  Conversion to Open Repair | 1
  Secondary Interventions | 18
  Aneurysm Enlargement | 5
  Clinically Significant Migration | 0
  Type IA Endoleak | 0
  Type IB Endoleak | 1
  Type IIIA Endoleak | 2
  Type IIIB Endoleak | 2
  Procedural Technical Success | 74

3. Secondary Outcome: Safety- Number of Major Adverse Events > 30 Days to 5 Years
Description: as for outcome 1
Time Frame: >30 Days to 5 Years
Population: All available data has been reported.
Measure: Number; unit: Number of events
Arm/Group | Ventana Fenestrated Stent Graft System
Number analyzed (Participants) | 74
Number of events
  All Cause Death | 28
  Bowel Ischemia | 2
  Myocardial Infarction | 3
  Paraplegia | 0
  Procedural Blood Loss | 0
  Renal Failure 1 - Temporary/Permanent Hemodialysis | 10
  Renal Failure 2 - Serum Creatinine >0.5mg/dL rise | 2
  Respiratory Failure 1 - Pneumonia | 9
  Respiratory Failure 2 - Ventilator >24 Hours | 3
  Stroke | 6

4. Secondary Outcome: Renal Dysfunction
Description: Renal Dysfunction is calculated at greater than 30% reduction starting at baseline
Time Frame: Discharge to 5 Years
Measure: Count of Participants; unit: Participants
Arm/Group | Ventana Fenestrated Stent Graft System
Number analyzed (Participants) | 76
Participants
  1-Month Follow-up | 9
  6-Month Follow-up | 11
  1-Year Follow-up | 22
  2-Year Follow-up | 16
  3-Year Follow-up | 11
  4-Year Follow-up | 11
  5-Year Follow-up | 8

5. Secondary Outcome: Endoleaks
Description: Endoleaks- Type IA, Type IB, Type II, Type IIIA, Type IIIB, Type IV, and Unknown Type
  Type I/III/IV Endoleak: Core Lab reported endoleak: between the endograft and the vessel either at the proximal attachment point (Type IA), or at the distal attachment point (Type IB), or between endograft components (Type III) or transgraft (Type IV).
  Type II Endoleak: Core Lab reported endoleak emanating from a patent collateral vessel (e.g., inferior mesenteric artery, lumbar artery).
Time Frame: 30 Days to 5 Years
Population: All available data based on different timepoints has been reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Ventana Fenestrated Stent Graft System
Number analyzed (Participants) | 69
Participants
  Type IA- 1 month | 0
  Type IB- 1 Month | 0
  Type II - 1 month | 11
  Type IIIA- 1 month | 0
  Type IIIB - 1 month | 0
  Type IV - 1 month | 0
  Unknown Type - 1 month | 6
  Type IA - 6 month: number analyzed (Participants) | 60
  Type IA - 6 month | 0
  Type IB- 6 Month: number analyzed (Participants) | 60
  Type IB- 6 Month | 0
  Type II- 6 Month: number analyzed (Participants) | 60
  Type II- 6 Month | 9
  Type IIIA- 6 Month: number analyzed (Participants) | 60
  Type IIIA- 6 Month | 0
  Type IIIB- 6 Month: number analyzed (Participants) | 60
  Type IIIB- 6 Month | 0
  Type IV- 6 Month: number analyzed (Participants) | 60
  Type IV- 6 Month | 0
  Unknown Type- 6 Month: number analyzed (Participants) | 60
  Unknown Type- 6 Month | 5
  Type IA- 1 Year: number analyzed (Participants) | 49
  Type IA- 1 Year | 0
  Type IB -1 Year: number analyzed (Participants) | 49
  Type IB -1 Year | 1
  Type II -1 Year: number analyzed (Participants) | 49
  Type II -1 Year | 6
  Type IIIA- 1 Year: number analyzed (Participants) | 49
  Type IIIA- 1 Year | 2
  Type IIIB- 1 Year: number analyzed (Participants) | 49
  Type IIIB- 1 Year | 2
  Type IV - 1 Year: number analyzed (Participants) | 49
  Type IV - 1 Year | 0
  Unknown Type- 1 Year: number analyzed (Participants) | 49
  Unknown Type- 1 Year | 4
  Type IA- 2 year: number analyzed (Participants) | 44
  Type IA- 2 year | 0
  Type IB- 2 Year: number analyzed (Participants) | 44
  Type IB- 2 Year | 0
  Type II- 2 Year: number analyzed (Participants) | 44
  Type II- 2 Year | 6
  Type IIIA- 2 Year: number analyzed (Participants) | 44
  Type IIIA- 2 Year | 2
  Type IIIB- 2 Year: number analyzed (Participants) | 44
  Type IIIB- 2 Year | 3
  Type IV- 2 Year: number analyzed (Participants) | 44
  Type IV- 2 Year | 0
  Unknown Type- 2 Year: number analyzed (Participants) | 44
  Unknown Type- 2 Year | 4
  Type IA- 3 Year: number analyzed (Participants) | 32
  Type IA- 3 Year | 0
  Type IB- 3 Year: number analyzed (Participants) | 32
  Type IB- 3 Year | 0
  Type II- 3 Year: number analyzed (Participants) | 32
  Type II- 3 Year | 5
  Type IIIA- 3 Year: number analyzed (Participants) | 32
  Type IIIA- 3 Year | 0
  Type IIIB- 3 Year: number analyzed (Participants) | 32
  Type IIIB- 3 Year | 1
  Type IV- 3 Year: number analyzed (Participants) | 32
  Type IV- 3 Year | 0
  Unknown Type- 3 Year: number analyzed (Participants) | 32
  Unknown Type- 3 Year | 2
  Type IA- 4 Year: number analyzed (Participants) | 22
  Type IA- 4 Year | 0
  Type IB- 4 Year: number analyzed (Participants) | 22
  Type IB- 4 Year | 0
  Type II- 4 Year: number analyzed (Participants) | 22
  Type II- 4 Year | 4
  Type IIIA- 4 Year: number analyzed (Participants) | 22
  Type IIIA- 4 Year | 0
  Type IIIB- 4 Year: number analyzed (Participants) | 22
  Type IIIB- 4 Year | 2
  Type IV- 4 Year: number analyzed (Participants) | 22
  Type IV- 4 Year | 0
  Unknown Type- 4 Year: number analyzed (Participants) | 22
  Unknown Type- 4 Year | 3
  Type IA- 5 Year: number analyzed (Participants) | 16
  Type IA- 5 Year | 0
  Type IB- 5 Year: number analyzed (Participants) | 16
  Type IB- 5 Year | 0
  Type II- 5 Year: number analyzed (Participants) | 16
  Type II- 5 Year | 1
  Type IIIA- 5 Year: number analyzed (Participants) | 16
  Type IIIA- 5 Year | 0
  Type IIIB- 5 Year: number analyzed (Participants) | 16
  Type IIIB- 5 Year | 1
  Type IV- 5 Year: number analyzed (Participants) | 16
  Type IV- 5 Year | 0
  Unknown Type- 5 Year: number analyzed (Participants) | 16
  Unknown Type- 5 Year | 2

6. Secondary Outcome: Clinical Utility Outcomes
Description: Clinical Utility Outcomes consist of: fluoroscopy time, Bifurcated device placement time, Renal Artery Cannulation time, F-EVAR time and total procedure time.
Time Frame: At the time of the procedure
Measure: Mean (Standard Deviation); unit: Mins
Arm/Group | Ventana Fenestrated Stent Graft System
Number analyzed (Participants) | 76
Mins
  Fluoroscopy Time | 58 (33)
  Bifurcated Device Placement Time | 56 (24)
  Renal Artery Cannulation Time | 35 (45)
  F-EVAR Time | 68 (32)
  Total Procedure Time | 205 (84)

7. Secondary Outcome: Time in ICU
Description: Number of days spent in the intensive care unit (ICU)
Time Frame: In-Hospital
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Ventana Fenestrated Stent Graft System
Number analyzed (Participants) | 76
Days | 3 (11)

8. Secondary Outcome: Time to Hospital Discharge
Description: Number of days from the index procedure to discharge from the hospital.
Time Frame: Hospital Discharge (Post-Procedure)
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Ventana Fenestrated Stent Graft System
Number analyzed (Participants) | 76
Days | 4 (8)

9. Secondary Outcome: Device Patency
Description: Device patency- Ventana & Bifurcated Occlusion, Left Renal Artery Occlusion, and Right Renal Artery Occlusion
Time Frame: 30 Days to 5 Years
Population: All available data at various timepoints have been reported
Measure: Count of Participants; unit: Participants
Arm/Group | Ventana Fenestrated Stent Graft System
Number analyzed (Participants) | 69
Participants
  Ventana & Bifurcated Occlusion - 1 Month | 0
  Left Renal Artery Occlusion - 1 month | 2
  Right Renal Artery Occlusion - 1month | 3
  Ventana & Bifurcated Occlusion- 6 Month: number analyzed (Participants) | 60
  Ventana & Bifurcated Occlusion- 6 Month | 0
  Left Renal Artery Occlusion- 6 Month: number analyzed (Participants) | 60
  Left Renal Artery Occlusion- 6 Month | 2
  Right Renal Artery Occlusion- 6 Month: number analyzed (Participants) | 60
  Right Renal Artery Occlusion- 6 Month | 2
  Ventana & Bifurcated Occlusion- 1 Year: number analyzed (Participants) | 49
  Ventana & Bifurcated Occlusion- 1 Year | 0
  Left Renal Artery Occlusion- 1 Year: number analyzed (Participants) | 49
  Left Renal Artery Occlusion- 1 Year | 2
  Right Renal Artery Occlusion- 1 Year: number analyzed (Participants) | 49
  Right Renal Artery Occlusion- 1 Year | 0
  Ventana & Bifurcated Occlusion- 2 Year: number analyzed (Participants) | 44
  Ventana & Bifurcated Occlusion- 2 Year | 0
  Left Renal Artery Occlusion- 2 Year: number analyzed (Participants) | 44
  Left Renal Artery Occlusion- 2 Year | 1
  Right Renal Artery Occlusion- 2 Year: number analyzed (Participants) | 44
  Right Renal Artery Occlusion- 2 Year | 1
  Ventana & Bifurcated Occlusion- 3 Year: number analyzed (Participants) | 32
  Ventana & Bifurcated Occlusion- 3 Year | 0
  Left Renal Artery Occlusion- 3 Year: number analyzed (Participants) | 32
  Left Renal Artery Occlusion- 3 Year | 0
  Right Renal Artery Occlusion- 3 Year: number analyzed (Participants) | 32
  Right Renal Artery Occlusion- 3 Year | 0
  Ventana & Bifurcated Occlusion - 4 Year: number analyzed (Participants) | 22
  Ventana & Bifurcated Occlusion - 4 Year | 0
  Left Renal Artery Occlusion- 4 Year: number analyzed (Participants) | 22
  Left Renal Artery Occlusion- 4 Year | 0
  Right Renal Artery Occlusion- 4 Year: number analyzed (Participants) | 22
  Right Renal Artery Occlusion- 4 Year | 0
  Ventana & Bifurcated Occlusion- 5 Year: number analyzed (Participants) | 16
  Ventana & Bifurcated Occlusion- 5 Year | 0
  Left Renal Artery Occlusion- 5 Year: number analyzed (Participants) | 16
  Left Renal Artery Occlusion- 5 Year | 0
  Right Renal Artery Occlusion- 5 Year: number analyzed (Participants) | 16
  Right Renal Artery Occlusion- 5 Year | 0

10. Secondary Outcome: Device Integrity
Description: Device Integrity- Device Migration, Ventana Stent Fracture, Left Renal Stent Fracture, Right Renal Stent Fracture, and Stent Kinking/ Compression
Time Frame: 30 Days to 5 Years
Population: All available data at various timepoints has been reported
Measure: Count of Participants; unit: Participants
Arm/Group | Ventana Fenestrated Stent Graft System
Number analyzed (Participants) | 73
Participants
  Device Migration- 6 Month: number analyzed (Participants) | 63
  Device Migration- 6 Month | 0
  Device Migration- 1 year: number analyzed (Participants) | 56
  Device Migration- 1 year | 0
  Device Migration- 2 year: number analyzed (Participants) | 48
  Device Migration- 2 year | 0
  Device Migration- 3 year: number analyzed (Participants) | 39
  Device Migration- 3 year | 0
  Device Migration- 4 year: number analyzed (Participants) | 28
  Device Migration- 4 year | 0
  Device Migration- 5 year: number analyzed (Participants) | 20
  Device Migration- 5 year | 0
  Ventana Stent Fracture- 1 Month: number analyzed (Participants) | 47
  Ventana Stent Fracture- 1 Month | 1
  Left Renal Stent Fracture- 1 Month: number analyzed (Participants) | 47
  Left Renal Stent Fracture- 1 Month | 1
  Right Renal Stent Fracture- 1 Month: number analyzed (Participants) | 47
  Right Renal Stent Fracture- 1 Month | 0
  Stent Kinking/ Compression- 1 Month | 0
  Ventana Stent Fracture- 6 Month: number analyzed (Participants) | 39
  Ventana Stent Fracture- 6 Month | 3
  Left Renal Stent Fracture- 6 Month: number analyzed (Participants) | 39
  Left Renal Stent Fracture- 6 Month | 2
  Right Renal Stent Fracture- 6 Month: number analyzed (Participants) | 39
  Right Renal Stent Fracture- 6 Month | 0
  Stent Kinking/ Compression- 6 Month: number analyzed (Participants) | 65
  Stent Kinking/ Compression- 6 Month | 0
  Ventana Stent Fracture- 1 Year: number analyzed (Participants) | 41
  Ventana Stent Fracture- 1 Year | 7
  Left Renal Stent Fracture- 1 Year: number analyzed (Participants) | 41
  Left Renal Stent Fracture- 1 Year | 7
  Right Renal Stent Fracture- 1 Year: number analyzed (Participants) | 41
  Right Renal Stent Fracture- 1 Year | 1
  Stent Kinking/ Compression- 1 Year: number analyzed (Participants) | 61
  Stent Kinking/ Compression- 1 Year | 0
  Ventana Stent Fracture- 2 Year: number analyzed (Participants) | 32
  Ventana Stent Fracture- 2 Year | 12
  Left Renal Stent Fracture- 2 Year: number analyzed (Participants) | 32
  Left Renal Stent Fracture- 2 Year | 8
  Right Renal Stent Fracture- 2 Year: number analyzed (Participants) | 32
  Right Renal Stent Fracture- 2 Year | 2
  Stent Kinking/ Compression- 2 Year: number analyzed (Participants) | 50
  Stent Kinking/ Compression- 2 Year | 0
  Ventana Stent Fracture- 3 Year: number analyzed (Participants) | 26
  Ventana Stent Fracture- 3 Year | 10
  Left Renal Stent Fracture- 3 Year: number analyzed (Participants) | 26
  Left Renal Stent Fracture- 3 Year | 5
  Right Renal Stent Fracture- 3 Year: number analyzed (Participants) | 26
  Right Renal Stent Fracture- 3 Year | 3
  Stent Kinking/ Compression- 3 Year: number analyzed (Participants) | 39
  Stent Kinking/ Compression- 3 Year | 0
  Ventana Stent Fracture- 4 Year: number analyzed (Participants) | 24
  Ventana Stent Fracture- 4 Year | 13
  Left Renal Stent Fracture- 4 Year: number analyzed (Participants) | 24
  Left Renal Stent Fracture- 4 Year | 3
  Right Renal Stent Fracture- 4 Year: number analyzed (Participants) | 24
  Right Renal Stent Fracture- 4 Year | 4
  Stent Kinking/ Compression- 4 Year: number analyzed (Participants) | 28
  Stent Kinking/ Compression- 4 Year | 0
  Ventana Stent Fracture- 5 Year: number analyzed (Participants) | 18
  Ventana Stent Fracture- 5 Year | 11
  Left Renal Stent Fracture- 5 Year: number analyzed (Participants) | 18
  Left Renal Stent Fracture- 5 Year | 3
  Right Renal Stent Fracture- 5 Year: number analyzed (Participants) | 18
  Right Renal Stent Fracture- 5 Year | 2
  Stent Kinking/ Compression- 5 Year: number analyzed (Participants) | 21
  Stent Kinking/ Compression- 5 Year | 0

11. Secondary Outcome: Aneurysm Sac Morphology
Description: Aneurysm Sac Morphology- Aneurysm Shape, Aneurysm Enlargement
Time Frame: 30 Days to 5 Years
Population: All available data has been reported
Measure: Count of Participants; unit: Participants
Arm/Group | Ventana Fenestrated Stent Graft System
Number analyzed (Participants) | 76
Participants
  Aneurysm Shape- Fusiform | 69
  Aneurysm Shape- Saccular | 7
  Aneurysm Enlargement - 6 months: number analyzed (Participants) | 63
  Aneurysm Enlargement - 6 months | 1
  Aneurysm Enlargement - 1 year: number analyzed (Participants) | 56
  Aneurysm Enlargement - 1 year | 4
  Aneurysm Enlargement - 2 year: number analyzed (Participants) | 48
  Aneurysm Enlargement - 2 year | 8
  Aneurysm Enlargement - 3 year: number analyzed (Participants) | 39
  Aneurysm Enlargement - 3 year | 8
  Aneurysm Enlargement - 4 year: number analyzed (Participants) | 28
  Aneurysm Enlargement - 4 year | 6
  Aneurysm Enlargement - 5 year: number analyzed (Participants) | 20
  Aneurysm Enlargement - 5 year | 6

12. Secondary Outcome: Aneurysm Sac Diameter
Description: Aneurysm Sac diameter changes
Time Frame: 30 Days to 5 Years
Population: All available data has been reported
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Ventana Fenestrated Stent Graft System
Number analyzed (Participants) | 76
mm
  Aneurysm Sac Diameter Changes - Screening / Baseline | 58.4 (7.9)
  Aneurysm Sac Diameter Changes - 1 month: number analyzed (Participants) | 73
  Aneurysm Sac Diameter Changes - 1 month | 59.3 (7.6)
  Aneurysm Sac Diameter Changes - 6 month: number analyzed (Participants) | 66
  Aneurysm Sac Diameter Changes - 6 month | 57.6 (7.4)
  Aneurysm Sac Diameter Changes - 1 year: number analyzed (Participants) | 61
  Aneurysm Sac Diameter Changes - 1 year | 57.1 (8.3)
  Aneurysm Sac Diameter Changes - 2 year: number analyzed (Participants) | 50
  Aneurysm Sac Diameter Changes - 2 year | 56.7 (8.2)
  Aneurysm Sac Diameter Changes - 3 year: number analyzed (Participants) | 39
  Aneurysm Sac Diameter Changes - 3 year | 55.5 (8.8)
  Aneurysm Sac Diameter Changes - 4 year: number analyzed (Participants) | 29
  Aneurysm Sac Diameter Changes - 4 year | 56.9 (10.4)
  Aneurysm Sac Diameter Changes - 5 year: number analyzed (Participants) | 21
  Aneurysm Sac Diameter Changes - 5 year | 59.7 (13.4)

13. Secondary Outcome: Clinical Utility Outcomes
Description: Clinical Utility Outcomes consists of: contrast volume and estimated blood loss.
Time Frame: At the time of the procedure
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Ventana Fenestrated Stent Graft System
Number analyzed (Participants) | 76
mL
  Contrast Volume | 132 (64)
  Blood loss | 401 (513)

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Ventana Fenestrated Stent Graft System
All-Cause Mortality (participants affected / at risk) | 30/76
Serious Adverse Events (participants affected / at risk) | 50/76
Other Adverse Events (participants affected / at risk) | 71/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ventana Fenestrated Stent Graft System (N=76)
Anemia (Blood and lymphatic system disorders) | 7 (7)
Hemorrhagic anemia (Blood and lymphatic system disorders) | 1 (1)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
AFib (Cardiac disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 3 (4)
Atrial fibrillation with rapid ventricular response (Cardiac disorders) | 2 (2)
Cardiac arrest (Cardiac disorders) | 2 (2)
Cardiogenic shock (Cardiac disorders) | 1 (1)
Cardiopulmonary arrest (Cardiac disorders) | 3 (3)
Congestive heart failure (Cardiac disorders) | 2 (2)
Coronary artery stenosis (Cardiac disorders) | 1 (1)
Heart block third degree (Cardiac disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 3 (3)
Non ST segment elevation myocardial infarction (Cardiac disorders) | 1 (1)
ST segment elevation myocardial infarction (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Ischemic optic neuropathy (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Acute pancreatitis (Gastrointestinal disorders) | 1 (2)
Bleeding gastrointestinal (Gastrointestinal disorders) | 1 (1)
Bowel ischemia (Gastrointestinal disorders) | 1 (1)
Bowel perforation (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Colitis ischemic (Gastrointestinal disorders) | 1 (1)
Diverticulosis (Gastrointestinal disorders) | 1 (1)
Emesis (Gastrointestinal disorders) | 1 (1)
GI bleed (Gastrointestinal disorders) | 1 (1)
Gastric ulcer perforation (Gastrointestinal disorders) | 1 (1)
Gastrointestinal bleed (Gastrointestinal disorders) | 2 (2)
Hemoperitoneum (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Inflammatory bowel disease (Gastrointestinal disorders) | 1 (1)
Left inguinal hernia (Gastrointestinal disorders) | 2 (2)
Mesenteric artery stenosis (Gastrointestinal disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 1 (1)
Necrotizing pancreatitis (Gastrointestinal disorders) | 1 (1)
Pancreatic duct obstruction (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Peptic ulcer disease (Gastrointestinal disorders) | 1 (1)
Peptic ulcer hemorrhage (Gastrointestinal disorders) | 1 (1)
Perforated gastric ulcer (Gastrointestinal disorders) | 1 (1)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1)
UGI bleed (Gastrointestinal disorders) | 2 (2)
Arterial stent occlusion (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Death (General disorders) | 4 (4)
Device fracture (General disorders) | 1 (1)
Device insertion difficult (General disorders) | 1 (1)
Device issue (General disorders) | 5 (5)
Device migration (General disorders) | 1 (1)
Edema (General disorders) | 1 (1)
Endoleak (General disorders) | 4 (5)
Fatigue aggravated (General disorders) | 1 (1)
Multi organ failure (General disorders) | 2 (2)
Stent malfunction (General disorders) | 3 (3)
Stent strut fracture (General disorders) | 4 (5)
Stent-graft angulation (General disorders) | 1 (1)
Stent-graft compression (General disorders) | 1 (1)
Stent-graft endoleak type IB (General disorders) | 1 (1)
Stent-graft endoleak type II (General disorders) | 2 (2)
Stent-graft endoleak type III (General disorders) | 5 (5)
Stent-graft malfunction (General disorders) | 1 (1)
Stent-graft material failure (General disorders) | 1 (1)
Vascular stent thrombosis (General disorders) | 1 (1)
Weakness (General disorders) | 2 (2)
Acute cholecystitis (Hepatobiliary disorders) | 1 (1)
Choledocholithiasis (Hepatobiliary disorders) | 1 (1)
Liver failure (Hepatobiliary disorders) | 1 (1)
Acute diverticulitis (Infections and infestations) | 1 (1)
Bacteremia (Infections and infestations) | 1 (1)
Chronic diverticulitis (Infections and infestations) | 1 (2)
Groin abscess (Infections and infestations) | 1 (1)
Incision site infection (Infections and infestations) | 2 (2)
Mycoplasma pneumoniae pneumonia (Infections and infestations) | 1 (1)
Nosocomial pneumonia (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 6 (9)
Postoperative wound infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Chronic subdural hematoma (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Fractured femur (excl neck) (Injury, poisoning and procedural complications) | 1 (1)
Fractured hip (Injury, poisoning and procedural complications) | 1 (1)
Graft complication (Injury, poisoning and procedural complications) | 2 (3)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1)
Hematuria traumatic (Injury, poisoning and procedural complications) | 1 (1)
In-stent arterial restenosis (Injury, poisoning and procedural complications) | 4 (4)
Injury to iliac artery (Injury, poisoning and procedural complications) | 2 (2)
Intraoperative bleeding (Injury, poisoning and procedural complications) | 1 (1)
Leg fracture (Injury, poisoning and procedural complications) | 1 (1)
Mental status changes postoperative (Injury, poisoning and procedural complications) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1)
Procedural bleeding (Injury, poisoning and procedural complications) | 3 (3)
Renal hematoma (Injury, poisoning and procedural complications) | 1 (1)
Scalp laceration (Injury, poisoning and procedural complications) | 1 (1)
Splenic hematoma (Injury, poisoning and procedural complications) | 1 (1)
Subdural hematoma (Injury, poisoning and procedural complications) | 2 (2)
Creatinine increased (Investigations) | 1 (1)
GFR decreased (Investigations) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1)
Gout flare (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Knee osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
weakness of Lower extremities (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis knee (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in hip (Musculoskeletal and connective tissue disorders) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Brain metastases (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thyroid carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Urothelial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Carotid artery stenosis (Nervous system disorders) | 2 (2)
Cerebral infarction (Nervous system disorders) | 1 (1)
Cerebral vascular disturbance (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Hemorrhagic transformation due to acute stroke (Nervous system disorders) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Intraventricular hemorrhage (Nervous system disorders) | 1 (1)
Progression of Alzheimer's disease (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Spinal cord ischemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Stroke (Nervous system disorders) | 2 (2)
Syncope (Nervous system disorders) | 2 (3)
Confusion (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1)
Acute kidney failure (Renal and urinary disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3)
Acute renal failure (Renal and urinary disorders) | 3 (3)
Acute tubular necrosis (Renal and urinary disorders) | 2 (2)
Bilateral renal artery stenosis (Renal and urinary disorders) | 4 (4)
Chronic renal failure (Renal and urinary disorders) | 2 (2)
Chronic renal failure worsened (Renal and urinary disorders) | 1 (1)
End stage renal disease (ESRD) (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Renal artery dissection (Renal and urinary disorders) | 1 (1)
Renal artery occlusion (Renal and urinary disorders) | 3 (4)
Renal artery stenosis (Renal and urinary disorders) | 13 (15)
Renal failure (Renal and urinary disorders) | 4 (4)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Renal parenchymal hemorrhage (Renal and urinary disorders) | 1 (1)
Unilateral renal artery stenosis (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Asphyxiation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung nodule (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Surgical intervention (Surgical and medical procedures) | 1 (1)
Umbilical hernia repair (Surgical and medical procedures) | 1 (1)
Abdominal aneurysm, ruptured (Vascular disorders) | 1 (1)
Abdominal aortic aneurysm enlargement (Vascular disorders) | 3 (3)
Aneurysm enlargement (Vascular disorders) | 1 (1)
Aortic aneurysm enlargement (Vascular disorders) | 1 (1)
Aortic aneurysm rupture (Vascular disorders) | 1 (1)
Arterial stenosis (Vascular disorders) | 2 (2)
Arterial thrombosis (Vascular disorders) | 1 (1)
Celiac artery occlusion (Vascular disorders) | 1 (1)
Critical limb ischemia (Vascular disorders) | 1 (1)
DVT (Vascular disorders) | 1 (1)
Femoral artery occlusion (Vascular disorders) | 1 (1)
Femoral artery stenosis (Vascular disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (2)
Hypertension (Vascular disorders) | 4 (4)
Hypotension (Vascular disorders) | 2 (2)
Hypovolemic shock (Vascular disorders) | 1 (1)
Arteriovenous Fistula placement (Vascular disorders) | 1 (1)
Iliac artery dissection (Vascular disorders) | 1 (1)
Iliac artery occlusion (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ventana Fenestrated Stent Graft System (N=76)
Anemia (Blood and lymphatic system disorders) | 10 (13)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 2 (3)
Splenic infarction (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3)
Acute heart failure (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 4 (4)
Atrial flutter (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Congestive heart failure (Cardiac disorders) | 1 (1)
Paroxysmal atrial fibrillation (Cardiac disorders) | 1 (1)
Premature atrial contraction (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Demand Ischemia (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 3 (3)
Uremic pericarditis (Cardiac disorders) | 1 (1)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1)
Hydrocele, unspecified (Congenital, familial and genetic disorders) | 1 (1)
Bilateral cataracts (Eye disorders) | 1 (1)
Blepharospasm (Eye disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 7 (7)
Bowel incontinence (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Constipation aggravated (Gastrointestinal disorders) | 2 (2)
Crohns disease aggravated (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (3)
Emesis (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 4 (4)
Localized intraabdominal fluid collection (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 9 (9)
Occlusion mesenteric artery (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Retroperitoneal hematoma (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (5)
Adverse drug reaction (General disorders) | 2 (2)
Chest pain (General disorders) | 3 (3)
Chest tightness (General disorders) | 1 (1)
Device migration (General disorders) | 1 (1)
Edema of lower extremities (General disorders) | 2 (3)
Endoleak (General disorders) | 4 (4)
Energy decreased (General disorders) | 1 (1)
Fever (General disorders) | 2 (2)
Leg edema (General disorders) | 1 (1)
Nodule (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 2 (3)
Rigors (General disorders) | 1 (1)
Stent malapposition (General disorders) | 1 (1)
Stent occlusion (General disorders) | 3 (3)
Stent strut fracture (General disorders) | 5 (5)
Stent-graft endoleak (General disorders) | 1 (1)
Stent-graft endoleak type IA (General disorders) | 1 (1)
Stent-graft endoleak type II (General disorders) | 6 (6)
Stent-graft endoleak type III (General disorders) | 1 (1)
Weakness (General disorders) | 3 (3)
Weakness generalised (General disorders) | 1 (1)
Left Arm Swelling (General disorders) | 1 (1)
Ear Wax build-up (General disorders) | 1 (1)
Liver cholestasis (Hepatobiliary disorders) | 1 (1)
Acute cystitis with hematuria (Hepatobiliary disorders) | 1 (1)
Acute bronchitis (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 3 (3)
C.difficile colitis (Infections and infestations) | 1 (1)
Candidemia (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 4 (5)
Clostridium difficile infection (Infections and infestations) | 1 (1)
Incision site cellulitis (Infections and infestations) | 1 (1)
Intestinal infection due to clostridium difficile (Infections and infestations) | 1 (1)
Left otitis externa (Infections and infestations) | 1 (1)
Methicillin-resistant staphylococcal aureus infection (Infections and infestations) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Pyelonephritis (Infections and infestations) | 1 (1)
Scrotal abscess (Infections and infestations) | 1 (1)
Tinea corporis (Infections and infestations) | 1 (1)
UTI (Infections and infestations) | 4 (4)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 6 (6)
Shingles (Infections and infestations) | 1 (1)
Anemia postoperative (Injury, poisoning and procedural complications) | 4 (4)
Ankle injury (Injury, poisoning and procedural complications) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Bruising of arm (Injury, poisoning and procedural complications) | 1 (1)
Confusion postoperative (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Contusion of knee (Injury, poisoning and procedural complications) | 1 (1)
Groin pain (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Hematoma postoperative (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
In-stent arterial restenosis (Injury, poisoning and procedural complications) | 1 (1)
Incision site erythema (Injury, poisoning and procedural complications) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 2 (2)
Injury to hand NOS (Injury, poisoning and procedural complications) | 1 (1)
Intraoperative bleeding (Injury, poisoning and procedural complications) | 1 (1)
Laceration of finger (Injury, poisoning and procedural complications) | 1 (1)
Laceration of leg (Injury, poisoning and procedural complications) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1)
Nausea postoperative (Injury, poisoning and procedural complications) | 1 (1)
Post procedural pain (Injury, poisoning and procedural complications) | 3 (3)
Postoperative bruise (Injury, poisoning and procedural complications) | 1 (1)
Postoperative pain (Injury, poisoning and procedural complications) | 7 (7)
Procedural bleeding (Injury, poisoning and procedural complications) | 3 (3)
Seroma (Injury, poisoning and procedural complications) | 6 (7)
Skull fracture NOS (Injury, poisoning and procedural complications) | 1 (1)
Splenic hematoma (Injury, poisoning and procedural complications) | 1 (1)
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 (1)
Vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Ankle brachial index decreased (Investigations) | 1 (1)
Blood creatinine decreased (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 6 (7)
Blood glucose increased (Investigations) | 1 (1)
Blood potassium increased (Investigations) | 1 (1)
Blood urea nitrogen increased (Investigations) | 1 (1)
Cardiac murmur (Investigations) | 1 (1)
Creatine kinase MB high (Investigations) | 1 (1)
Creatine kinase increased (Investigations) | 1 (1)
Creatinine blood increased (Investigations) | 3 (3)
Creatinine increased (Investigations) | 2 (2)
Decreased hemoglobin (Investigations) | 1 (1)
Hematocrit decreased (Investigations) | 1 (1)
Hematocrit low (Investigations) | 1 (1)
Hemoglobin low (Investigations) | 1 (1)
Increased serum creatinine (Investigations) | 3 (3)
Magnesium low (Investigations) | 1 (1)
Mean arterial pressure increased (Investigations) | 1 (1)
Potassium increased (Investigations) | 1 (1)
Raised INR (Investigations) | 1 (2)
Raised WBC (Investigations) | 1 (1)
Sodium decreased (Investigations) | 1 (1)
Systolic murmur (Investigations) | 1 (1)
TSH decrease (Investigations) | 1 (1)
Urine output decreased (Investigations) | 2 (2)
WBC increased (Investigations) | 1 (1)
Weight loss (Investigations) | 2 (2)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1)
Hyperammonemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 4 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 2 (2)
Acute back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Axillary lump (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Calf pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Cervical spine degeneration (Musculoskeletal and connective tissue disorders) | 1 (1)
Cervicalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Chronic back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cramp in hand (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Foot Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Hematoma muscle (Musculoskeletal and connective tissue disorders) | 1 (1)
Knee pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Leg pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Low back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Lower extremities weakness of (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1)
Rotator cuff tendinitis (Metabolism and nutrition disorders) | 1 (1)
Skin tear (Musculoskeletal and connective tissue disorders) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1)
Weakness of arms (Musculoskeletal and connective tissue disorders) | 1 (1)
Lung neoplasm NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Aneurysm cerebral (Nervous system disorders) | 1 (1)
Clonus (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 6 (7)
Headache post-traumatic (Nervous system disorders) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1)
Lightheadedness (Nervous system disorders) | 1 (1)
Nerve pain (Nervous system disorders) | 2 (2)
Neuropathy (Nervous system disorders) | 1 (1)
Numbness in hand (Nervous system disorders) | 1 (1)
Paresthesia lower limb (Nervous system disorders) | 1 (1)
Parkinsonism (Nervous system disorders) | 1 (1)
Positional dizziness (Nervous system disorders) | 1 (1)
Restless leg syndrome (Nervous system disorders) | 1 (1)
Sensory polyneuropathy axonal (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Stent-graft endoleak (Product Issues) | 1 (1)
Cocaine abuse (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Depression worsened (Psychiatric disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 3 (3)
Mood disorder NOS (Psychiatric disorders) | 1 (1)
Sleep disorder (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Acute on chronic renal failure (Renal and urinary disorders) | 1 (1)
Acute renal failure (Renal and urinary disorders) | 2 (2)
Acute renal insufficiency (Renal and urinary disorders) | 2 (2)
Atrophy kidney (Renal and urinary disorders) | 2 (2)
Bladder hypertrophy (Renal and urinary disorders) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Creatinine abnormal NOS (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (2)
Impaired renal function (Renal and urinary disorders) | 1 (1)
Kidney stone (Renal and urinary disorders) | 1 (1)
Renal artery occlusion (Renal and urinary disorders) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 1 (1)
Renal cyst (Renal and urinary disorders) | 1 (1)
Renal infarct (Renal and urinary disorders) | 1 (1)
Renal infarction (Renal and urinary disorders) | 1 (1)
Uremia (Renal and urinary disorders) | 1 (1)
Urethral spasm (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 6 (7)
Penile bleed (Renal and urinary disorders) | 1 (1)
Breast inflammation (Reproductive system and breast disorders) | 1 (1)
Cervical cyst (Reproductive system and breast disorders) | 1 (1)
Scrotal edema (Reproductive system and breast disorders) | 1 (1)
Scrotal swelling (Reproductive system and breast disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3 (4)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung mass (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Lung nodule (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pleural plaque (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Singers nodules (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 3 (3)
Itching (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (4)
Rash both legs (Skin and subcutaneous tissue disorders) | 1 (1)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin disorder NOS (Skin and subcutaneous tissue disorders) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 2 (2)
Skin rash (Skin and subcutaneous tissue disorders) | 1 (1)
Skin red (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Arterial repair NOS (Surgical and medical procedures) | 1 (1)
Abdominal aortic aneurysm enlargement (Vascular disorders) | 1 (2)
Aneurysm enlargement (Vascular disorders) | 1 (1)
Claudication (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2)
Essential hypertension (Vascular disorders) | 1 (2)
Femoral artery dissection (Vascular disorders) | 1 (1)
Hematoma (Vascular disorders) | 2 (3)
Hypertension (Vascular disorders) | 8 (9)
Hypertension aggravated (Vascular disorders) | 4 (4)
Hypertension exacerbated (Vascular disorders) | 1 (1)
Hypertension worsened (Vascular disorders) | 2 (2)
Hypertensive crisis (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 7 (7)
Iliac artery aneurysm (Vascular disorders) | 1 (1)
Iliac artery dissection (Vascular disorders) | 1 (1)
Leg ischemia (Vascular disorders) | 1 (1)
Lymphocele (Vascular disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Raynauds (Vascular disorders) | 1 (1)
Refractory hypertension (Vascular disorders) | 1 (1)
Vasovagal episode (Vascular disorders) | 1 (1)
Venous insufficiency (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-02-27): https://cdn.clinicaltrials.gov/large-docs/45/NCT01491945/Prot_SAP_000.pdf
  • Informed Consent Form (2012-02-07): https://cdn.clinicaltrials.gov/large-docs/45/NCT01491945/ICF_001.pdf